CLINICAL TRIAL: NCT02129868
Title: An Open-label, Single-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy and Safety of a Novel Automated Overnight Closed-loop Glucose Control System on Day 1 of Continuous Glucose Monitoring Sensor Insertion in Comparison to Day 3 to 4 After Sensor Insertion in Children and Adolescents With Type 1 Diabetes
Brief Title: Automated Closed-loop in Children and Adolescents With Type 1 Diabetes
Acronym: APCam09
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Director of Research, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APCam09
Record Dates: First submitted 2014-04-23; First posted 2014-05-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases; Autoimmune Diseases
Keywords: Type 1 diabetes; Closed-loop glucose control; Artificial Pancreas; Continuous subcutaneous insulin infusion; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed-loop on day 1 of CGM sensor life (Experimental): Glucose level is controlled by the automated closed-loop glucose control system on day 1 after CGM sensor insertion.
  Interventions: Device: Closed-loop (Android Closed-Loop platform)
- Closed-loop on day 3 of CGM sensor life (Active Comparator): Glucose level is controlled by the automated closed-loop glucose control system on day 3 or 4 after CGM sensor insertion.
  Interventions: Device: Closed-loop (Android Closed-Loop platform)

INTERVENTIONS:
Device: Closed-loop (Android Closed-Loop platform) — The closed-loop system is purpose-built and comprises a hand-held computer containing a model predictive control (MPC) based glucose control algorithm and communicating with the CGM device and the insulin pump.
  The Android Closed-Loop platform employs the Medtronic MiniMed Paradigm® Veo™ insulin pump system with CGM capability (use of MiniLink™Transmitter and sensor). A Radiofrequency (RF) translator module translates the RF protocol to Bluetooth® technology. An Android device containing an algorithm will use sensor glucose data to calculate pump strokes.

SUMMARY:
People with type 1 diabetes need regular insulin injections or continuous delivery of insulin using a pump. Keeping blood sugars in the normal range is known to reduce long term complications. However, achieving treatment goals can be very difficult due to the risk of low glucose levels (hypoglycaemia). One solution is to use a system where the amount of insulin injected closely matches the blood sugar levels on a continuous basis. This can be achieved by what is known as a "closed loop system" where a small glucose sensor placed under the skin communicates with a computer containing an algorithm that drives a subcutaneous insulin pump. Previous studies conducted under carefully controlled clinical research facility environment, in Cambridge, United Kingdom, as well as several other centres have shown that closed-loop glucose control is superior to usual insulin pump therapy. The next logical step in the development pathway is to test closed loop systems in the home environment. An essential requirement for conducting closed-loop studies outside clinical research facility is an automated system where wireless data transmission takes place between the glucose sensor and insulin pump.

The purpose of the present study is to evaluate the efficacy and safety of automated overnight closed-loop, in children and adolescents with type 1 diabetes, using a novel system which has greatest potential for use in the home setting. The study will take place at a clinical research facility on two occasions, using a standardised protocol. The performance of the closed-loop system will be evaluated on day 1 of continuous glucose monitoring (CGM) sensor life as compared to on days 3 to 4 of sensor life. Data and experience gained from this study will be used for further refinements and development of the system for future home use.

DETAILED DESCRIPTION:
The main objective of the current study is to evaluate the efficacy, safety and utility/reliability of a novel automated overnight closed-loop glucose control system in children and adolescents with type 1 diabetes. This will inform the future development of closed-loop systems in children and adolescents aged 6 to 18 years with type 1 diabetes.

This is an open-label, randomised, 2-period cross-over study, using the Medtronic Android closed loop platform or similar, comparing the safety and efficacy of overnight closed loop glucose control on day 1 compared with day 3 to 4 of CGM sensor life. Participants will be randomised to undergo two overnight studies in a clinical research facility, during which glucose levels will be controlled by the computer-based closed-loop algorithm on day 1 of CGM sensor insertion or day 3 to 4 after sensor insertion.

A total of 16 children and adolescents with T1D between 6 and 18 years of age will be recruited through the Outpatient Diabetes Clinic in the Department of Paediatrics, Addenbrooke's Hospital and Paediatric Diabetes Centres in London, Norwich, and Ipswich, to allow for 12 available for assessment. All participants will be on insulin pump treatment with a good knowledge of insulin dose adjustments. The study will take place at the Wellcome Trust Clinical Research Facility (WTCRF), Cambridge. Participants will be admitted at the clinical research facility in the evening and stay until the following morning. During the two closed-loop visits, automated closed-loop glucose control with wireless data transmission will be performed. A Model-Predictive-Control algorithm will determine the insulin infusion rate based on interstitial glucose measured by a continuous subcutaneous glucose monitoring (CGM) system. Intravenous sampling for glucose and insulin levels will also be carried out on both study visits for post hoc validation of glucose sensor data and for future modelling purposes.

The primary efficacy endpoint is the time spent in the target plasma glucose range from 3.9 to 8 mmol/L. Safety evaluation is focused on the frequency and duration of episodes of hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 6 and 18 years of age.
* The subject has had type 1 diabetes, as defined by WHO criteria for at least 1 year or is confirmed C-peptide negative.
* The subject will have been an insulin pump user for at least 3 months, with a good knowledge of insulin dose adjustment.
* HbA1c between below 11 % based on analysis from central laboratory.
* The subject is literate in English.
* The subject is willing to undertake all study related activities.

Exclusion Criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease.
* Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results.
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids, non-selective beta-blockers and MAO inhibitors.
* Known or suspected allergy against insulin.
* Subjects with clinically significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
* Patient is pregnant, or breast feeding during the period of the study.
* Total daily insulin dose ≥ 2 Units/kg/day
* Total daily insulin dose < 10 Units/day
* Severe visual impairment
* Severe hearing impairment
* Subjects using implanted internal pacemaker

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time spent with plasma glucose concentration in the target glucose range from 3.9 to 8.0 mmol/l. | 10 hours
  The primary outcome measure is time spent with plasma glucose concentration in the target range (3.9-8.0mmol/L) between 21:30 on Day 1 and 07:30 on Day 2 (10 hours), as obtained with closed-loop insulin delivery on day 1 of CGM sensor insertion as compared with closed-loop insulin delivery on day 3 to 4 of CGM sensor insertion.

SECONDARY OUTCOMES:
Time spent with plasma glucose concentration below the target range (<3.9mmol/L) between 21:30 on Day 1 and 07:30 on Day 2 (10 hours). | 10 hours
Time spent with plasma glucose concentration above the target range (>8mmol/L) between 21:30 on Day 1 and 07:30 on Day 2 (10 hours). | 10 hours
Mean and standard deviation of plasma glucose levels between 21:30 on Day 1 and 07:30 on Day 2 (10 hours). | 10 hours
Total insulin delivery between 21:30 on Day 1 and 07:30 on Day 2 (10 hours). | 10 hours
Total basal insulin delivery between 21:30 on Day 1 and 07:30 on Day 2 (10 hours). | 10 hours
Plasma insulin concentrations between 21:30 on Day 1 and 07:30 on Day 2 (10 hours). | 10 hours
Absolute relative difference between matched pairs of subcutaneous glucose sensor and reference plasma glucose. | 10 hours

OTHER OUTCOMES:
Percentage of time the system is functioning as intended in active closed-loop mode. | 14 hours
  Reliability / utility evaluation
CGM failure (defined as no CGM glucose available for whatever reason; failure rate ) | 14 hours
  Reliability / utility evaluation
Problems with user interface / Android platform (failure rate) | 14 hours
  Reliability / utility evaluation
Loss of communication between different system components (failure rate) | 14 hours
  Reliability / utility evaluation
number of episodes of hypoglycaemia (plasma glucose ≤ 3.5mmol/l) | 14 hours
  Safety Evaluation
number of episodes of hypoglycaemia (plasma glucose ≤ 2.8mmol/l) | 14 hours
  Safety evaluation
number of subjects experiencing hypoglycaemia | 14 hours
  Safety evaluation
nature and severity of any other adverse events | 14 hours
  Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357
- [Background] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665
- [Background] Elleri D, Allen JM, Biagioni M, Kumareswaran K, Leelarathna L, Caldwell K, Nodale M, Wilinska ME, Acerini CL, Dunger DB, Hovorka R. Evaluation of a portable ambulatory prototype for automated overnight closed-loop insulin delivery in young people with type 1 diabetes. Pediatr Diabetes. 2012 Sep;13(6):449-53. doi: 10.1111/j.1399-5448.2012.00903.x. Epub 2012 Jul 23. PMID 22817340
- [Background] Kumareswaran K, Elleri D, Allen JM, Harris J, Xing D, Kollman C, Nodale M, Murphy HR, Amiel SA, Heller SR, Wilinska ME, Acerini CL, Evans ML, Dunger DB, Hovorka R. Meta-analysis of overnight closed-loop randomized studies in children and adults with type 1 diabetes: the Cambridge cohort. J Diabetes Sci Technol. 2011 Nov 1;5(6):1352-62. doi: 10.1177/193229681100500606. PMID 22226252
- [Result] Tauschmann M, Allen JM, Wilinska ME, Ruan Y, Thabit H, Acerini CL, Dunger DB, Hovorka R. Sensor Life and Overnight Closed Loop: A Randomized Clinical Trial. J Diabetes Sci Technol. 2017 May;11(3):513-521. doi: 10.1177/1932296816678631. Epub 2016 Nov 11. PMID 27837162